CLINICAL TRIAL: NCT07158060
Title: The Effects of Breathing Exercises on Exam Anxiety, Attention Deficit, and Academic Achievement in Students Preparing for University Entrance Exams
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Minel YILDIRIM, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-74555795-050.04-1394112; E-74555795-050.04-1394112 (Other: Istanbul University-Cerrahpasa)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Academic Acheivement; Attention; Exam Anxiety; Breathing Exercises; Students
Keywords: Breathing Exercises; Exam Anxiety; Attention; Academic Achievement; Students; High School Seniors
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two parallel groups. The intervention group will practice structured breathing exercises, while the control group will continue their usual study routine. The intervention will last for 8 weeks with two sessions per week. Baseline characteristics such as age, gender, and academic performance will be balanced between groups to ensure comparability.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises Group (Intervention) (Experimental): Participants in this group will practice structured breathing exercises designed to reduce exam anxiety and improve attention and academic performance. The intervention consists of 8 weeks of training, with two sessions per week. Techniques include diaphragmatic breathing, the 4-7-8 method, and Nadi Shodhana (alternate nostril breathing). Participants are encouraged to practice daily at home using instructional materials provided.
  Interventions: Behavioral: Breathing Exercises
- Control Group (Usual Study Routine) (No Intervention): Participants in this group will continue their normal study activities without any additional breathing exercises or structured interventions. They will follow their standard academic schedule throughout the 8-week study period.

INTERVENTIONS:
Behavioral: Breathing Exercises — Breathing Exercises This intervention
  Arms: Breathing Exercises Group (Intervention)

SUMMARY:
This study investigates the effects of breathing exercises on exam anxiety, attention, and academic achievement in students preparing for university entrance exams. University entrance exams are significant milestones in students' educational and career paths, often causing high levels of stress and anxiety. These psychological pressures can negatively impact learning, focus, and overall academic performance.

The study will involve students who volunteer to participate and meet the inclusion criteria. Participants will be guided through structured breathing exercises designed to reduce stress and enhance concentration. The program will be conducted over several sessions, during which students will practice specific breathing techniques under supervision.

Primary outcomes of the study include the assessment of changes in exam anxiety levels, attention, and academic performance. Secondary outcomes may include students' self-reported stress management skills and overall well-being. Data will be collected using validated questionnaires, attention tests, and academic performance records.

The purpose of this research is to determine whether regular practice of targeted breathing exercises can provide practical benefits for students, helping them manage anxiety, improve focus, and achieve better academic outcomes. Findings from this study may also offer guidance for educators, parents, and healthcare providers on effective, low-cost interventions to support students during high-pressure academic periods.

Participants are encouraged to follow instructions carefully and attend all sessions to gain the full benefit of the intervention. Participation is voluntary, and students can withdraw at any time without any negative consequences. Confidentiality of all collected data will be strictly maintained.

By contributing to this research, participants will help advance understanding of non-pharmacological methods to improve student mental health and academic performance, potentially shaping future educational and stress-management programs.

DETAILED DESCRIPTION:
Breathing, the process of inhalation and exhalation, is a vital physiological function for human life. The respiratory system facilitates the intake of oxygen and the removal of carbon dioxide. Oxygen obtained through respiration supports numerous essential bodily functions, including energy production, cellular activity, acid-base balance, and brain health. In children, respiratory physiology exhibits differences compared to adults, influenced by anatomical and physiological characteristics that change with age. As children grow, these differences gradually diminish. During adolescence, the growth rate of organs and systems increases significantly.

According to the World Health Organization, adolescence is a unique developmental stage between childhood and adulthood, crucial for establishing the foundations of lifelong health. Adolescents undergo rapid physical, cognitive, and psychosocial development, which influences their emotions, thought processes, decision-making, and interactions with the world. These interactions also impact academic achievement.

The process of preparing for university entrance examinations can be a stressful and anxiety-inducing period for many students. Common sources of anxiety include social and parental expectations, time management challenges, and career uncertainty. Methods for managing anxiety include participation in social activities, hobbies, meditation, and breathing exercises. Modern education emphasizes not only cognitive skill development but also the enhancement of emotional and social abilities. Supporting students in attention, stress coping, and anxiety management, especially in high-pressure situations like exams, is directly related to academic success. Accordingly, incorporating attention-enhancing practices, breathing techniques, or mindfulness-based interventions into educational programs is recommended. In a study by Işık (2022), mindfulness and attention training provided to primary school students resulted in significant improvements in Bourdon Attention Test scores, suggesting that combining cognitive attention training with psychological relaxation techniques can be effective.

Nursing encompasses more than physical care; it adopts a holistic approach that addresses mental and emotional well-being. School nurses and other healthcare professionals within educational settings play a crucial role in supporting students' psychological well-being, monitoring exam-related anxiety, and providing early intervention if necessary. Literature indicates that nurses actively guiding students in attention and stress management programs significantly reduce anxiety levels. Furthermore, nurses can support the application of psycho-educational methods, such as breathing exercises, relaxation techniques, and mindfulness practices, while monitoring students' attention levels.

Breathing exercises involve conscious control of respiration to achieve relaxation, reduce stress, increase energy, and improve overall health. Various techniques provide distinct benefits, with controlled breathing serving as the initial step in promoting physical and mental relaxation. These exercises are particularly effective in alleviating physiological tension, such as nausea, tremors, or shortness of breath. Physiologically, controlled breathing activates the parasympathetic nervous system and reduces cortisol levels, producing a calming effect on the body. It is suggested that approximately 20 minutes of breathing exercises are required to allow the body to achieve a relaxed and focused state after stress onset. Practicing breathing exercises 10-15 minutes before exams may help prevent the physiological manifestations of anxiety.

The relationship between breathing exercises and stress management is well-documented and widely accepted in modern psychology and medicine. Historically, breathing practices have been used in various cultures. In ancient India, Pranayama, a key component of yoga, involved conscious breath control to regulate life energy (prana) for mental clarity, energy enhancement, and meditation practice. In ancient Greece and Rome, Stoics considered breath control essential for mental clarity and emotional balance. During the Middle Ages and Renaissance, Sufi breathing exercises, including dhikr (repetition of divine names), were employed for spiritual development. In the modern era, yoga practices and mindfulness meditation techniques, which incorporate breath awareness and control, have become widely adopted for stress management and mental health improvement.

Commonly used breathing techniques include:

Diaphragmatic Breathing (Abdominal Breathing): Deep breathing involving expansion and contraction of the abdomen, promoting relaxation and efficient oxygen intake.

4-7-8 Technique: Inhale for 4 seconds, hold for 7 seconds, exhale for 8 seconds, calming the nervous system.

Nadi Shodhana (Alternate Nostril Breathing): Alternating inhalation and exhalation through each nostril to balance energy flow and promote mental calmness.

Breathing exercises can be applied during exam preparation, during exams, and after exams to enhance learning, attention, memory, focus, and organizational skills. These techniques are not limited to academic stress but can be used in daily life to improve well-being. Practical applications include managing intense exam anxiety, difficulty concentrating, memory recall issues, post-exam uncertainty, mental fatigue, and stress reduction during high-pressure periods.

Scientific evidence demonstrates that regular practice of breathing exercises reduces stress and anxiety, enhances focus, improves physical health, promotes emotional balance, and increases sleep quality. Studies on students show that such practices can positively influence attention, anxiety management, and cognitive performance, ultimately supporting better academic outcomes.

Despite their potential benefits, few studies have investigated the use of breathing exercises as a holistic school-based intervention for students preparing for university entrance exams. Consequently, this study is designed to evaluate the effects of structured breathing exercises on exam anxiety, attention deficit, and academic achievement in high school senior students. The findings are expected to contribute to the literature and provide evidence-based recommendations for educational and nursing interventions.

ELIGIBILITY:
Inclusion Criteria:

* 12th grade students
* Obtaining consent from both parents and students
* No language, hearing, intellectual, or psychological disabilities
* Able to speak and understand Turkish
* Planning to take the university entrance exam
* Voluntary participation in the study
* Selecting two high schools with similar entrance scores for the study
* Students with high scores on the Westside Test Anxiety Scale

Exclusion Criteria:

* Presence of any chronic disease
* Presence of any heart disease
* Currently using any psychiatric medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Attention Levels | 8 months
  Students' attention levels will be assessed using the Bourdon Attention Test or a similar standardized attention assessment tool. The change in attention scores from baseline to post-intervention will be evaluated.
Exam Anxiety | 8 Months
  The level of exam-related anxiety will be assessed using the Westside Test Anxiety Scale (WTAS). This scale ranges from 1 to 5, with higher scores indicating greater levels of test anxiety. Higher scores reflect higher levels of exam anxiety, while lower scores reflect lower levels. Although no fixed cut-off point exists, when applied to larger groups, students scoring +1 standard deviation and above may be considered as having high exam anxiety, whereas those scoring -1 standard deviation and below may be considered as having low exam anxiety. The primary outcome is the change in anxiety scores from baseline to post-intervention.
Academic Achievement | 8 months
  Academic performance will be measured using students' exam scores or school grades. Scores range from 0 to 100, with higher scores indicating better academic achievement. The change in academic achievement from baseline to post-intervention will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Minel YILDIRIM, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided